CLINICAL TRIAL: NCT05202106
Title: Digital Support Systems to Improve Child Health and Development in Peru - a Randomized Controlled Trial
Brief Title: Digital Support Systems to Improve Child Health and Development in Peru
Acronym: DigitalECD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Harvard University (Other); ETH Zurich (Switzerland) (Other); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DigitalECD
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Child Development
Keywords: child development; stimulation; mobile phones; digital interventions
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Intervention Model Description: This study is designed as an open-label, 3-arm parallel trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment, and final data analysis will be conducted using de-identified and blinded data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Families in the control group will not receive any interventions and will simply complete baseline and endline surveys.
- Home visits (Experimental): Families in the home visiting arm will receive visits by trained child development agents every two weeks between enrollment and 2 years of age.
  Interventions: Behavioral: Home visits
- Afini (Experimental): Families in the Afini arm will be introduced to the Afini app on Messenger and encouraged to use this platform throughout the study.
  Interventions: Other: Afini App

INTERVENTIONS:
Behavioral: Home visits — Home visits entail a visit a children's home every two weeks. During this visit, trained child development agents will engage parents in activities with the child and provide basic toys and learning materials.
  Arms: Home visits
Other: Afini App — Afini is an app designed to help parents provide nurturing environments and stimulation to their young children. Most caregivers currently connect to the platform via Facebook Messenger; once they sign up, the platforms start engaging the caregiver by recommending age-specific health- and development-promoting activities. Rather than just hoping that caregivers will later engage in these activities, the virtual assistant directly observes whether caregivers access the materials for the recommended activity, and asks caregivers to provide feedback on each task.
  Arms: Afini

SUMMARY:
About 250 million children under age five are at risk of not reaching their developmental potential due to continued exposure to ill health, malnutrition and lack of appropriate learning environments. A large number of initiatives have been launched in recent years to support early childhood development, with home visiting programs increasingly being recognized as a key strategy for improving child wellbeing. However, the most effective ways to reach families in low income settings remain unclear due to the large expense associated with personal family visits. This project assesses the effectiveness and equity of a newly developed digital platform designed to deliver evidence-based, individualized parenting support through automated services. The Afinidata platform uses state-of-the art machine learning algorithms to allow caregivers to get answers to questions about child health and development, while also identifying and promoting age- and development-appropriate activities for parents to support their children. The goal of this study is to rigorously assess the reach, impact and cost effectiveness of this digital platform in a poor rural population through a randomized controlled trial. The study is designed as mixed-methods evaluation approach with repeated feedback into the Afinidata system. A total of 2400 newborns will be enrolled in a randomized controlled trial in San Marcos, Peru, and followed up for two years. The primary study outcome will be children's healthy development at 24 months of age assessed through the Bayley Scales of Infant and Toddler Development (BSID-III). Secondary outcomes will be systems utilization, program coverage and cost-effectiveness, as well as caregiver satisfaction. If proven effective, this innovative digital platform may increase global access to low-cost parental support -a widely recognized key strategy for improving child well-being.

DETAILED DESCRIPTION:
Children in low and middle income countries continue to be exposed to large amount of adversity, undermining their health and early development. While a large number of programs have been launched recently to support children in their home environment, the best ways to reach families in low income settings remain unclear.

In this study we will assess the impact of a newly developed virtual platform designed to support parents of young children in low resource settings. The Afinidata platform was launched in 2017 to support caregivers online via social media messengers that are now almost universally used in low and middle income countries. The Afinidata platform allows caregivers to get answers to questions about child health and development, while also identifying and promoting age- and development-appropriate activities for parents to support their children.

The main objective of this study is to assess the reach, impact, cost-effectiveness and scalability of the Afinidata platform for improving early childhood health and development. The primary study outcomes will be children's overall development at age 2, assessed through Global Scales for Early Development (GSED) long form. Secondary outcomes will include parental engagement as well as children's motor, cognitive, language and socio-emotional development.

A total of 164 communities in San Marcos, Cajabamba and Cajamarca provinces will be identified for the trial, and divided into 3 groups: a control group (72 community clusters, 1080 caregiver-child dyads) a home visiting group (20 community clusters, 300 caregiver-child dyads), and an online intervention group using the Afinidata platform (72 community clusters, 1080 caregiver-child dyads).

All 2400 caregivers in the trials, as well as 240 children participating in the national Cuna Mas program (external reference group) will be visited in their homes for a baseline interview at the beginning and an end-line interview at the end of the study.

Caregivers in the home visiting group will receive a home visit by a trained agent every two weeks following the guidelines of the nationally developed CUNA MAS program starting from six months of age until the child turns 2.

Caregivers in the Afinidata group will be visited once in the beginning of the study and introduced to the online system. After this initial visit, caregivers will be supported through the Afinidata platform. A randomly selected subgroup of Afinidata users (20 clusters) will also receive small biweekly or monthly data transfers of about USD 2 to support access to Afini's data systems.

ELIGIBILITY:
Inclusion Criteria:

* children residing in the study area

Exclusion Criteria:

* children with disabilities
* families planning to leave study area
* families participating in national Cuna Mas program

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Child Development at age 2 years | 2 years
  The primary study outcome will be overall child development as measured by the Global Scales for Early Development (GSED). Total scores on the GSED scales will be converted to z-scores for the analysis. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Caregiver mental health and stress | 2 years after enrollment (child age 2)
  Caregiver mental health and stress scores will be assessed using the Depression, Anxiety and Stress Scales (DASS). The scale contains three subscores for depression, stress and anxiety - higher scores on these scales indicate mental health problems (worse outcomes)
Caregiver self-efficacy | 2 years after enrollment
  Caregiver self-efficacy will be assessed at endline - when child turn 2 years. Higher scores on this scale indicate better outcomes.
Home stimulation | Endline - 2 years after enrollment
  Home stimulation measures caregiver engagement with children. We will measure this using the MICS home stimulation questionnaire. This scale ranges from 0-6 - higher scores imply more home stimulation (better outcomes).
Caregiver screen time | Endline - 2 years after enrollment
  Caregiver screen time will be collected at endline through a (self-reported) question to caregivers.

CONTACTS AND LOCATIONS:
Locations (2):
- Cayetano Heredia University, Lima, Peru
- Swiss Tropical and Public Health Institute, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The trial data will be made publicly available after publication of the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After publication

REFERENCES:
- [Derived] Hartinger Pena SM, Mausezahl D, Jaggi L, Aguilar L, Alvarado Llatance M, Castellanos A, Huaylinos Bustamante ML, Hinckley K, Charles McCoy D, Zhang C, Fink G. Digital Support Systems to Improve Child Health and Development in Peru: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 14;12:e50371. doi: 10.2196/50371. PMID 38096020